CLINICAL TRIAL: NCT04826523
Title: Venetoclax (Venclexta Tablet) Post-Marketing Surveillance for AML Patients
Brief Title: Study of Oral Venetoclax Tablets to Evaluate Adverse Events and Change in Disease Activity in Participants Above 19 Years of Age With Acute Myeloid Leukemia (AML)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-444
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML); AML; Venetoclax; Venclexta; Venclyxto; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with Venetoclax: Participants who were prescribed venetoclax for the treatment of Acute Myeloid Leukemia (AML) will be enrolled for this study.

SUMMARY:
Acute Myeloid Leukemia (AML) is an aggressive and rare cancer of myeloid cells (a white blood cell responsible for fighting infections). This study will assess how safe and effective oral venetoclax is in participants with AML . Adverse events and change in disease activity will be monitored under routine clinical practice.

Venetoclax is an approved drug for treatment of Acute Myeloid Leukemia (AML). Around 600 participants of age 19 years and above will be enrolled in the study in multiple medical institutions across South Korea.

Participants will receive oral venetoclax tablets as prescribed by their physician in the routine clinical practice. Participants will be observed for 7 cycles ( each cycle is 28 days).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

--Acute Myeloid Leukemia (AML) participants who have been prescribed oral Venetoclax tablets for the first time according to the approved label.

Exclusion Criteria:

* Participants with contraindications to Venetoclax as listed on the approved local label.
* Participants receiving Venetoclax in clinical trials.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Myeloid Leukemia (AML) participants who are prescribed Venetoclax within the approved label shall be enrolled in the study according to the clinical judgment of the physician in charge of the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Reported Serious Adverse Event/Drug Reaction | 32 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants who Achieved Complete Remission (CR) | 28 weeks
  The percentage of participants with complete remission (CR) will be calculated based on the modified International Working Group (IWG) criteria for AML.
Percentage of Participants who Achieved Complete Remission With Incomplete Hematologic Recovery (CRi) | 28 weeks
  Incomplete regeneration of bone marrow (CRi) as defined in the study protocol.
The Percentage of Participants who Achieved Composite Complete Remission (CR+CRi) | 28 weeks
  Composite Complete Remission (CRc) is defined as Complete Remission (CR) + CRi (CR with incomplete blood count recovery) based on protocol.
Median Time to Achieve Complete Remission [CR] (month) | 28 weeks
  Time from date of first oral Venetoclax intake and the date of the assessment having documented Complete Remission (in months).
Median Time to Achieve CRi | 28 weeks
  Time from the date of first oral venetoclax intake and the date of the assessment having documented Complete Remission with incomplete Hematologic recovery (CRi).
Median Overall Survival [OS] (month) | 28 weeks
  Time from the date of first oral venetoclax intake to the date of death from any cause.
Median Progression Free Survival [PFS] (month) | 28 weeks
  Median time to achieve Progression Free Survival (PFS) which is the time from [enrollment or randomization or first dose] to disease progression or death [to the first occurrence of radiographic progression determined by blinded independent central review or death from any cause], whichever occurs first.
Overall Response Rate (ORR) Based on Effectiveness Outcome | 28 weeks
  Overall Response Rate (ORR) is the proportion of the responders to the total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- South Korea (10):
  - Pusan National University Hospital /ID# 239010, Busan, Busan Gwang Yeogsi
  - Kosin University Gospel Hospital /ID# 257399, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 257398, Daegu, Daegu Gwang Yeogsi
  - Gachon University Gil Medical Center /ID# 239008, Incheon, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 257478, Hwasun-gun, Jeonranamdo
  - Korea University Anam Hospital /ID# 231022, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 257477, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 239009, Seoul, Seoul Teugbyeolsi
  - Yeungnam University Medical Center /ID# 239007, Daegu
  - Yonsei University Health System Severance Hospital /ID# 239006, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/